Statistical Analysis Plan: Solid Tumor Studies

Version 1.0 dated: 30 January 2018

Protocol Numbers: ACE-ST-003, ACE-ST-005, ACE-ST-006, ACE-ST-007, ACE-ST-208

Title: A Master Statistical Analysis Plan for Solid Tumor Studies

Version: 1.0

Version date: 30 January 2018

The undersigned have reviewed and approved this plan



#### CONFIDENTIAL

This document (and all copies thereof) is the property of Acerta Pharma and contains valuable trade secrets and confidential information, including proprietary technical and business information. By accepting this document, you agree that the Confidential Information contained herein will not be disclosed to others without prior written authorization from Acerta Pharma and shall only be used for the purposes intended by the document.

Statistical Analysis Plan: Solid Tumor Studies


## A Master Statistical Analysis Plan for

# Solid Tumor Studies including ST-003, ST-005, ST-006, ST-007, and ST-208

Version: Version 1.0 Date: 30Jan 2018

Studies Statistician:

Acerta Pharma 

Statistical Analysis Plan: Solid Tumor Studies


Table 1. A List of Applicable Studies Covered by This SAP

| Protocol<br>Number | Treatment groups | Indication | Phase | Protocol Title |
|---|---|---|---|---|
| ACE-ST-003 | Acalabrutinib<br>vs<br>Acalabrutinib +<br>Pembrolizumab | Pancreatic<br>Cancer | 2 | A Phase 2 Proof-of-Concept<br>Study of ACP-196 Alone and<br>in Combination with<br>Pembrolizumab in Subjects<br>with Advanced or Metastatic<br>Pancreatic Cancer |
| ACE-ST-005 | Pembrolizumab<br>vs<br>Acalabrutinib +<br>Pembrolizumab | Bladder Cancer | 2 | Randomized Phase 2 Trial of ACP-196 and Pembrolizumab Immunotherapy Dual CHECKpoint Inhibition in Platinum Resistant Metastatic Urothelial Carcinoma |
| ACE-ST-006 | Pembrolizumab<br>vs<br>Acalabrutinib +<br>Pembrolizumab | Head and Neck<br>Cancer | 2 | A Phase 2 Proof-of-Concept<br>Study of the Combination of<br>ACP-196 and Pembrolizumab<br>in Subjects with Advanced<br>Head and Neck Squamous<br>Cell Carcinoma |
| ACE-ST-007 | Pembrolizumab<br>vs<br>Acalabrutinib +<br>Pembrolizumab | Non-small Cell<br>Lung Cancer | 2 | A Phase 2 Proof-of Concept<br>Study of the Combination of<br>ACP-196 and Pembrolizumab<br>in Subjects with Advanced<br>Non-small Cell Lung<br>Carcinoma |
| ACE-ST-208 | Acalabrutinib<br>vs<br>Acalabrutinib +<br>Pembrolizumab | Ovarian Cancer | 2 | A Phase 2 Proof-of-Concept<br>Study of ACP-196 Alone and<br>in Combination with<br>Pembrolizumab in Subjects<br>with Recurrent Ovarian Cancer |

Acerta Pharma 

Statistical Analysis Plan: Solid Tumor Studies


#### **TABLE OF CONTENTS**

| Table | e of C | ontents. | | 3 |
|---|---|---|---|---|
| Table | e of A | bbreviati | ons | 5 |
| 1. | INTE | RODUCT | ION | 7 |
| 2. | OBJI<br>2.1<br>2.2<br>2.3 | Primary<br>Second | S | 7<br>7 |
| 3. | STUI<br>3.1<br>3.2 | Study D | RVIEW<br>Design Size | 8 |
| 4. | STUI<br>4.1<br>4.2<br>4.3 | Safety E<br>Efficacy | POINTS Endpoints Endpoints tory Endpoints | 9<br>9 |
| 5. | HYP | OTHESE | ES AND MULTIPLICITY | 9 |
| 6. | ANA<br>6.1<br>6.2<br>6.3 | Safety A<br>Efficacy | ETSAnalysis Set<br>Evaluable Analysis Setacokinetic/Pharmacodynamic Analyses Set | 10<br>10 |
| 7. | FINA | L ANAL | YSIS AND CLINICAL STUDY REPORT | 10 |
| 8. | STA <sup>-</sup><br>8.1<br>8.2<br>8.3<br>8.4<br>8.5 | General<br>Subject<br>Importa<br>Demogr | L METHODS OF ANALYSIS I Principles Accountability nt Protocol Deviations raphic and Baseline Characteristics ent and Medications Prior Anticancer Regimens Concomitant Medications Exposure to Investigational Product | 10<br>11<br>11<br>11<br>11 |
| | 8.6 | Safety A<br>8.6.1<br>8.6.2<br>8.6.3<br>8.6.4<br>8.6.5 | Analyses Adverse Events Adverse Events of Clinical Interest Laboratory Test Results Vital Signs ECOG Performance Status | 12<br>13<br>13 |

| | 8.7 | Efficac | y Analyses | 13 |
|---|---|---|---|---|
| | | 8.7.1 | Best Overall Response, Disease Control Rate and Overall Response Rate | 13 |
| | | 8.7.2 | Duration of Response | |
| | | 8.7.3 | Progression-free Survival | 14 |
| | | 8.7.4 | Overall Survival | 15 |
| | | 8.7.5 | Serum Cancer Antigens CA-19-9 and CA-125 | 15 |
| | | 8.7.6 | Exploratory Efficacy Endpoints | 15 |
| | | 8.7.7 | Other Exploratory Efficacy Endpoints | 16 |
| | | 8.7.8 | Pharmacokinetic, Pharmacodynamic and Biomarker | |
| | | | Analyses | |
| | 8.8 | Sensiti | ivity Analyses | 16 |
| 9. | CHA | NGES I | FROM PROTOCOL-SPECIFIED ANALYSES | 16 |
| 10. | LITE | RATUR | RE CITATIONS / REFERENCES | 17 |
| 11. | APP | ENDICE | ≣S | 18 |
| | | | ions | |
| | | | ation Rules for Partial or Missing Dates | |
| | | | ring Rules for Progression-free Survival | |
| | | | ring Rules for Overall Survival | |
| | | | s of Clinical Interest for acalabrutinib | |
| | | | of Clinical Interest for a combination of acalabrutinib and | |
| | | pembr | olizumab | 24 |

Statistical Analysis Plan: Solid Tumor Studies


#### TABLE OF ABBREVIATIONS

AE adverse event

ALT alanine aminotransferase
AST aspartate aminotransferase

BID twice per day
BMI Body mass index
BOR best overall response

CA19-9 cancer antigen 19-9 (carbohydrate antigen 19-9)

CI confidence interval
CR complete response
CRF case report form
CSR clinical study report

CTCAE Common Terminology Criteria for Adverse Events

DCR disease control rate
DLT dose-limiting toxicity
DOR duration of response

ECOG Eastern Cooperative Oncology Group

FDA Food and Drug Administration

HNSCC head and neck squamous cell carcinoma

ICF informed consent form

IPD Important Protocol Deviation

ir immune-related

irRECIST immune-related response criteria

IV intravenous or intravenously

MDSCs myeloid-derived suppressor cells

MedDRA Medical Dictionary for Regulatory Activities

NCI National Cancer Institute

NSCLC non-small cell lung cancer

ORR overall response rate

OS overall survival
PD pharmacodynamics
PD progressive disease

PD-L1 programmed death ligand-1 PFS progression-free survival

PK pharmacokinetics

PO orally

PR partial response Q3W every 3 weeks

RECIST Response Evaluation Criteria in Solid Tumors

SAE serious adverse event SAP statistical analysis plan

Statistical Analysis Plan: Solid Tumor Studies


SD stable disease SOC system organ class

TEAE treatment-emergent adverse event

ULN upper limit of normal

WHODRUG World Health Organization WHO Drug Dictionary

Statistical Analysis Plan: Solid Tumor Studies


#### 1. INTRODUCTION

The purpose of this statistical analysis plan (SAP) is to provide details of the statistical analyses that have been outlined within the protocols of including ST-003(pancreatic cancer), ST-005 (bladder cancer), ST-006 (head and neck squamous cell carcinoma, HNSCC), ST-007 (non-small cell lung cancer, NSCLC), and ST-208 (ovarian cancer). The scope of this plan includes the final analysis. Any changes to the methods described in this SAP will be documented in each clinical study report (CSR).

#### 2. OBJECTIVES

#### 2.1 **Primary Objective**

- To characterize the safety profile of acalabrutinib and pembrolizumab in subjects with solid tumors in each of the five studies including ST-003 (pancreatic cancer), ST-005 (bladder cancer), ST-006 (HNSCC), ST-007 (NSCLC), and ST-208 (ovarian cancer).
- To determine the best overall response rate and overall response rate (ORR)
  of pembrolizumab monotherapy and the combination of acalabrutinib and
  pembrolizumab. This applies to ST-005, ST-006 and ST-007.

#### 2.2 Secondary Objective

- To evaluate the efficacy (multiple efficacy endpoints including ORR, PFS and OS) of acalabrutinib monotherapy and acalabrutinib and pembrolizumab combination treatment in subjects with solid tumors using standard response criteria. This applies to ST-003 and ST-208.
- To determine progression-free survival (PFS) in subjects treated with pembrolizumab monotherapy and the combination of acalabrutinib and pembrolizumab. This applies to ST-005, ST-006, and ST-007.
- To evaluate the overall survival (OS) in subjects treated with pembrolizumab monotherapy and the combination of acalabrutinib and pembrolizumab. This applies to ST-005, ST-006, and ST-007.



Acerta Pharma 

Statistical Analysis Plan: Solid Tumor Studies




#### 3. STUDY OVERVIEW

#### 3.1 Study Design

These five studies are phase 2, multicenter, open-label, randomized studies evaluating acalabrutinib or pembrolizumab monotherapy and the combination of acalabrutinib and pembrolizumab in subjects with solid tumors. Subjects meeting the eligibility criteria for the study will be randomized 1:1 to one of the following arms:

<u>Arm 1:</u> Acalabrutinib 100 mg administered orally (PO) twice per day (BID) (ST-003, ST-208) **or** Pembrolizumab 200 mg administered as an intravenous (IV) infusion every 3 weeks (Q3W) (ST-005, ST-006, ST-007)

Arm 2: Acalabrutinib 100 mg PO BID plus Pembrolizumab 200 mg IV Q3W Acalabrutinib treatment can continue for subjects who are tolerating therapy and not progressing. Pembrolizumab study treatment is for 24 months from the date of first dose for subjects who are tolerating therapy and not progressing. Subjects who have confirmed progressive disease on the combination of pembrolizumab and acalabrutinib will discontinue study treatment. Subjects who have confirmed progressive disease on monotherapy arm may start combination until a second disease progression. Disease progression will be determined based on irRECIST guidelines. Also pembrolizumab treatment can end for subjects with confirmed complete response (CR) if treatment has been administered for at least 24 weeks and 2 doses of pembrolizumab have been administered after confirmation of CR.

Refer to Protocol section 3 for more details.

#### 3.2 Sample Size

The planned sample sizes per arm for each of the studies are listed below. For sample size justification, reference corresponding study protocols:

| Study Arm 1: Acalabrutinib Arm 1: Pembrolizuma | | Arm 1: Pembrolizumab | Arm 2: Acalabrutinib |
|---|---|---|---|
| Study | Alli I. Acaiabiutiilib | Ami i. Pembionzumab | + Pembrolizumab |
| ST-003 | 38 | | 38 |
| ST-005 | | 37 | 37 |
| ST-006 | | 37 | 37 |

Acerta Pharma 

Statistical Analysis Plan: Solid Tumor Studies


| ST-007 | | 37 | 37 |
|--------|----|----|----|
| ST-208 | 38 | | 38 |

#### 4. STUDY ENDPOINTS

#### 4.1 Safety Endpoints

Type, frequency, severity, timing of onset, duration, and relationship to either
or both study drug of any treatment-emergent adverse events (TEAEs) or
abnormalities of laboratory tests, serious adverse events (SAEs), AEs leading
to dose modification, dose delay and discontinuation of any study drug

#### 4.2 Efficacy Endpoints

- Disease control rate (DCR) defined as stable disease (SD), partial response (PR) or CR based on modified RECIST 1.1 criteria. DCR by RECIST will be considered the primary endpoint of ST-003
- ORR, defined as PR or CR based on modified RECIST 1.1 criteria. ORR by RECIST will be considered the primary endpoint of ST-005, ST-006, ST-007, and ST-208
- Duration of response (DOR)
- PFS
- OS
- Change in serum cancer antigen CA-19-9. This applies to ST-003 only
- Change in serum cancer antigen CA-125. This applies to ST-208 only



#### 5. HYPOTHESES AND MULTIPLICITY

This series of solid tumor studies are proof of concept studies. No formal hypothesis will be tested and no multiplicity adjustments will be made.

Acerta Pharma 

Statistical Analysis Plan: Solid Tumor Studies


#### 6. ANALYSIS SETS

The following definitions will be used for the efficacy and safety analysis populations.

#### 6.1 Safety Analysis Set

The safety analysis set includes all subjects who receive at least one dose of any study drug (either acalabrutinib or pembrolizumab). The safety analysis set will be used for evaluating the safety and efficacy endpoints with the exception of DOR. The analyses of DOR will be conducted on the subset of the safety analysis set who achieve CR or PR as their best overall response.

#### 6.2 Efficacy Evaluable Analysis Set

All subjects in the safety analysis set who have ≥ 1 evaluable response assessment after the first dose of study drug (either acalabrutinib or pembrolizumab). Sensitivity analyses of efficacy endpoints will be carried out on the efficacy-evaluable population.

#### 6.3 Pharmacokinetic/Pharmacodynamic Analyses Set

Pharmacokinetic/Pharmacodynamic evaluable analysis set will be defined by PK/PD group.

#### 7. FINAL ANALYSIS AND CLINICAL STUDY REPORT

Planned final analysis will be conducted once last subject exits study and database is locked. The CSR will be written based on the final analysis.

#### 8. STATISTICAL METHODS OF ANALYSIS

#### 8.1 General Principles

Descriptive statistics [including means, standard deviations, medians, minimum and maximum for continuous variables and frequency, proportions and confidence intervals (CIs) for discrete variables] will be used to summarize data as appropriate.

Calculation of time to event or duration of event endpoints will be based on the study day of the event or censoring date rather than visit number or visit label. Missing efficacy or safety data will not be imputed unless otherwise specified.

The following rules will be used for the days to months/years conversion:

- 1 month= 30.4375 days;
- 1 year= 365.25 days.

Statistical Analysis Plan: Solid Tumor Studies


All summaries will be presented by treatment group.

#### 8.2 Subject Accountability

The number of subjects enrolled by site will be presented. Subject disposition will be summarized for all enrolled subjects including the following information:

- Proportion of subjects who received study drug
- Proportion of subjects with study drug discontinuation and primary reason for study drug discontinuation
- Proportion of subjects discontinuing study and reasons for study discontinuation
- Time on study

#### 8.3 Important Protocol Deviations

Important Protocol Deviations (IPDs) categories are defined and managed by the study team during the IPD reviews throughout the study before database lock. The final IPD list for each study is used to produce the summary of IPDs and the listing of subjects with IPDs, respectively.

#### 8.4 Demographic and Baseline Characteristics

Summaries of demographic characteristics will be presented for age, age category (< 65, ≥ 65), gender, race, ethnicity, and geographic region for each study.

Baseline characteristics will be presented for Eastern Cooperative Oncology Group (ECOG) performance status, disease stage, tumor grade where relevant, number of prior anticancer therapies for each study.

#### 8.5 Treatment and Medications

#### 8.5.1 Prior Anticancer Regimens

Summary statistics will be presented for prior anticancer regimens (might include multiple therapies) and prior cancer-related surgery for each study. Prior cancer therapy categories will be adjudicated by the medical monitor.

#### 8.5.2 Concomitant Medications

Concomitant medications will be coded and tabulated according to the World Health Organization Drug Dictionary (WHODRUG).

Statistical Analysis Plan: Solid Tumor Studies


#### 8.5.3 Exposure to Investigational Product

Number of subjects who received at least one dose of acalabrutinib, pembrolizumab or both, duration of exposure, average daily dose of acalabrutinib, average dose of pembrolizumab per administration cycle, and relative dose intensity will be summarized for each investigational product and by treatment group.

Exposure parameters are defined in more detail in Appendix 12.1.

#### 8.6 Safety Analyses

#### 8.6.1 Adverse Events

The Medical Dictionary for Regulatory Activities (MedDRA v20.1 or higher) will be used to code all AEs to a system organ class and a preferred term. The severity of the AE will be assessed by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03. Study drug-related AEs are those assessed by investigator as related.

All AE tables will be summarized by original treatment group and crossover group for each study. For subjects who crossed-over from monotherapy to a combination therapy of acalabrutinib and pembrolizumab, AEs experienced up to crossover date will summarized under monotherapy arm, while AEs on or after the cross-over date (1st dose date of second study drug added) will be summarized under crossover group.

TEAEs are defined as those events that occur or worsen on or after the first dose of study drug, through the treatment phase, and within 30 days following the last dose of acalabrutinib or within 90 days following the last dose of pembrolizumab.

TEAEs will be summarized by system organ class (SOC) and preferred terms in descending order of frequency, by CTCAE toxicity grade. Drug-related TEAEs, serious TEAEs, TEAEs leading to treatment discontinuation and removal from study will be summarized by SOC and preferred terms as well as by preferred teams only in descending order of frequency and by CTCAE toxicity grade.

Death information is reported in the study exit case report form (CRF) for all deaths. Incidences of deaths are to be reported, along with the primary cause of death.

Acerta Pharma 

Statistical Analysis Plan: Solid Tumor Studies


#### 8.6.2 Adverse Events of Clinical Interest

Events of Clinical Interest identified for acalabrutinib and combination of acalabrutinib with pembrolizumab will be summarized for each study. The definitions of these categories are part of Appendix 12.5 and 12.6.

#### 8.6.3 Laboratory Test Results

Laboratory data up to 30 days after last dose or the safety follow-up visit date, whichever is later, will be reported in SI units. Applicable laboratory results will be graded according to CTCAE Version 4.03. For each laboratory parameter, the baseline laboratory value/grade is defined as the last laboratory value/grade collected on or prior to the date of the first dose of study drug. Treatment-emergent laboratory abnormalities for selected parameters will be summarized.

#### 8.6.4 Vital Signs

Body temperature, heart rate (beats/min), systolic blood pressure (mmHg), diastolic blood pressure (mmHg), respiratory rate (breaths/min), and weight will be collected for each study as scheduled in protocol Appendix. For each parameter, summary statistics (mean, standard deviation, median, and range) will be produced for baseline, maximum, and minimum value.

#### 8.6.5 ECOG Performance Status

ECOG performance status scores will be summarized for each treatment group using shift table. The shifts in scores from baseline to worst ECOG score on treatment will be summarized.

#### 8.7 Efficacy Analyses

### 8.7.1 Best Overall Response, Disease Control Rate and Overall Response Rate

DCR is defined as the proportion of subjects who achieve a best response of SD, PR or CR at any point of the study. The primary endpoint for ST-003 is DCR by RECIST1.1 criteria by investigators.

ORR is defined as the proportion of subjects who achieve a best response of PR or CR at any point of the study. The primary endpoint for ST-005, ST-006, ST-007, and ST-208 is ORR by RECIST1.1 criteria by investigators.

Acerta Pharma 

Statistical Analysis Plan: Solid Tumor Studies


The primary analysis of DCR and ORR will be conducted using safety analysis set. DCR and ORR will be calculated with the corresponding exact binomial 2-sided 95% CI for each original treatment arm and separately for subjects who crossed over from a monotherapy to a combination therapy. Monotherapy subjects who crossed-over will be summarized according to their original treatment assignment up to the point of crossover, and then summarized as a crossover subject using their response immediately prior to crossover as a new baseline for their combination treatment. A sensitivity analysis using efficacy evaluable analysis set will also be presented.

Descriptive statistics will be provided for best overall response for each treatment group. The number and proportion of subjects within each category of response will be presented.

#### 8.7.2 Duration of Response

The DOR is defined as the interval from the first documentation of response to the earlier of the first documentation of definitive disease progression or death from any cause. The DOR will only be summarized for subjects in safety analysis set who achieved response (CR or PR) at any point of the study. Kaplan-Meier methods will be used to estimate event-free curves and corresponding quantiles (including the median).

For crossover subjects who originally started on monotherapy, the DOR will only be summarized/listed if ORR for this group is non-zero. If confirmed response is achieved after the crossover, the DOR for a combination therapy will be summarized.

Data from surviving, non-progressing subjects will be censored at the date of the last adequate disease assessment that is on or before the start date of the new antitumor therapy. Data from subjects who have disease progression or die after more than one missed visit will be censored at the last visit date before the missing assessments which lack objective disease assessment. The details of definition of progression events and censoring rules are the same as for PFS endpoint and are listed in Appendix 12.3.

#### 8.7.3 Progression-free Survival

Progression-free survival is defined as the interval from the start of therapy to the earlier of the first documentation of objective disease progression or death from any cause. Kaplan-Meier methods will be used to estimate the event-free curves and corresponding quantiles (including the median).

Acerta Pharma 

Statistical Analysis Plan: Solid Tumor Studies


For crossover subjects who originally started on monotherapy, the PFS will only be summarized/listed if ORR for this group is non-zero.

Data from surviving, non-progressing subjects will be censored at the date of the last adequate disease assessment that is on or before the start date of the new antitumor therapy. Data from subjects who have disease progression or die after more than one missed visit will be censored at the last visit date prior to the missing assessments which lack objective disease assessment. The details of definition of progression events and censoring rules for primary and sensitivity analyses of PFS are listed in Appendix 12.3.

In the primary analysis using safety analysis set, study treatment end date will be used as the date of progression for subjects who discontinued study treatment due to disease progression or death prior to 1<sup>st</sup> radiographic assessment. Data for subjects who discontinued study treatment prior to 1<sup>st</sup> radiographic assessment due to reasons other than disease progression or death will be censored at their study treatment start date.

#### 8.7.4 Overall Survival

Overall survival is defined as the time from treatment start date until date of death due to any cause. Subjects who are known to be alive or whose survival status is unknown will be censored at the date last known to be alive. Subjects who lost to follow-up for survival immediately after randomization will be censored at first dose date (Appendix 12.4). OS will be summarized for safety analysis set only and based on original treatment assignment. Crossover subjects who originally started on monotherapy and cross over to a combination treatment will be summarized as part of the original monotherapy group for OS. The analysis methods for OS will be similar to those described for PFS.

#### 8.7.5 Serum Cancer Antigens CA-19-9 and CA-125

Changes in CA-19-9 (ST-003) and CA-125 (ST-208) will be evaluated using descriptive statistics using safety analysis set.

#### 8.7.6 Exploratory Efficacy Endpoints

In addition to evaluation of DCR, ORR, DOR and PFS by RECIST 1.1 criteria exploratory endpoints of irDCR, irORR, irDOR and irPFS were planned to be evaluated by irRECIST criteria (Appendix 7 or 8 in the protocols). For studies that did not collect these immune-related responses no analysis will be performed.

Acerta Pharma 

Statistical Analysis Plan: Solid Tumor Studies


#### 8.7.7 Other Exploratory Efficacy Endpoints

Time to initial response (PR or better) in months will be calculated and summarized.

#### 8.7.8 Pharmacokinetic, Pharmacodynamic and Biomarker Analyses

Additional pharmacodynamic, pharmacokinetic and biomarker analyses may be performed, as deemed appropriate. A separate analysis plan for these analyses will be developed by PK/PD group.

#### 8.8 Sensitivity Analyses

Sensitivity analyses will be done using efficacy evaluable analysis set for efficacy endpoints of ORR. if the primary and sensitivity analysis of ORR are consistent, we won't perform sensitivity analysis using efficacy evaluable analysis set for DOR, PFS, and OS. They are also referenced in corresponding parts of section 9.7.

#### 9. CHANGES FROM PROTOCOL-SPECIFIED ANALYSES

Exploratory endpoints of irDCR, irORR, irDOR and irPFS were planned to be evaluated by irRECIST criteria. For studies that did not collect these endpoints no analysis will be performed. These changes will also be documented in the Clinical Study Report.

Also, one event of clinical interest (ECIs) defined in these protocols (overdose) will not be applicable for this final analysis. Instead, an expanded list of ECIs will be summarized based on the emerging clinical data for acalabrutinib and recent FDA submission in MCL. Overdose, if occurred, will be summarized as part of the important protocol deviations.

Acerta Pharma 

Statistical Analysis Plan: Solid Tumor Studies


#### 10. LITERATURE CITATIONS / REFERENCES

 Guidance for Industry. Clinical Trail Endpoints for the Approval of Cancer Drugs and Biologics. FDA. May 2007. <a href="http://www.fda.gov/downloads/Drugs/GuidanceComplianceRegulatoryInformation/Guidances/ucm071590.pdf">http://www.fda.gov/downloads/Drugs/GuidanceComplianceRegulatoryInformation/Guidances/ucm071590.pdf</a>

- 2. Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0, USDHHS, NIH, NCI; publish date May 28, 2009 (v4.03: June 14, 2010).
- 3. Eisenhauer EA, Therasse P, Bogaerts J, et al. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer 2009;45:228-247.
- 4. Bohnsack O, Ludajic K, Hoos A. Adaption of the immune-related response criteria: irRECIST. EMSO 2014, Abstract 4958.

Acerta Pharma 

Statistical Analysis Plan: Solid Tumor Studies


#### 11. APPENDICES

#### 12.1 Definitions

#### Study Day

The study day will be calculated in reference to the first dose date of study drug. Study Day 1 is defined as the first dose date of study drug. For assessments that occur on or after the first dose date of study drug, study day is defined as (date of assessment – first dose date of study drug + 1). For assessments that occur prior to the first dose date of study drug, study day is defined as (date of assessment – first dose date of study drug). There is no Study Day 0.

#### **Duration of Exposure**

The duration of exposure to acalabrutinib or pembrolizumab will be calculated in months as (last dose date - first dose date + 1) / 30.4375. The gaps in treatment will be included. The duration of exposure in days will be used for planned dose calculation.

#### **Total Dose**

Total dose received is a sum of all actual doses taken through the treatment duration and will be presented in grams. For scheduled drug administration visits that are skipped the actual dose will be 0.

#### Average Daily Dose (Acalabrutinib)

Average daily dose is total dose divided by duration of exposure in days.

#### Average Dose per administration cycle (Pembrolizumab)

Average dose <u>per administration cycle</u> is total dose divided by number of cycles for pembrolizumab study treatment.

#### Relative Dose Intensity

Relative dose intensity is the ratio of total dose to the protocol-specified total dose through the duration of exposure.

Acerta Pharma 

Statistical Analysis Plan: Solid Tumor Studies


#### 12.2 Imputation Rules for Partial or Missing Dates

Imputation of partial dates will be made for AE onset and stop dates, start and end dates of concomitant medication, start date of subsequent anticancer therapy, date of initial diagnosis and death date. If dates are completely missing, no imputation will be made. For any partial date with missing year, no imputation will be made.

The general rule for imputation is:

- If only day is missing, then the 15<sup>th</sup> of the month will be used.
- If only year is present, then June 30<sup>th</sup> will be used.

If such imputation date for initial diagnosis is on or after date of first dose, then date of first dose – 1 will be used. If such imputed date for subsequent anticancer therapies is before date of last dose, then date of last dose + 1 will be used.

If the imputed date is for an AE start date and is in the same year and month as but before the first dose date, then the first dose date will be used, or if the imputed AE start date is after the AE end date, then the AE end date will be used. If the imputed date is for an AE start date and is in the same year and month as but after the last dose date + 30 days, then the last dose date + 30 days will be used.

If the imputed date is for an AE end date and is after the death date, then the death date will be used, or if the imputed AE end date is before the AE start date, then the AE start date will be used.

Every effort will be made to obtain complete dates for deaths. If both month and day are missing for death date or a death date is totally missing, do not impute and censor the subject survival time. If death year and month are available but day is missing, the following algorithm will be used:

- If mmyyyy for last contact date = mmyyyy for death date, set death date to the day after the last contact date.
- If mmyyyy for last contact date < mmyyyy for death date, set death date to the first day of the death month.
- If mmyyyy for last contact date > mmyyyy for death date, data error and do not impute.

Acerta Pharma 

Statistical Analysis Plan: Solid Tumor Studies


#### 12.3 Censoring Rules for Progression-free Survival

| Situation | PFS1 | |
|---|---|---|
| | Date of Progression or<br>Censoring | Outcome |
| Progression documented on scheduled visit | Date of scheduled visit | Progression |
| Progression documented between scheduled visits | Date of unscheduled visit | Progression |
| Treatment discontinuation for undocumented progression | Date of last visit with adequate assessment | Censor |
| Death before first PD assessment | Date of death | Progression |
| Death between adequate assessment visits | Date of death | Progression |
| Death or progression after only one missed visit | Date of death | Progression |
| Death or progression after 2 or more missed visits | Date of last visit with adequate assessment | Censor |
| Death or progression after 2 or <u>more missed</u> visits and only <u>baseline</u> tumor assessment available | Date of 1st dose of study drug | Censor |
| No baseline tumor assessments | Date of 1st dose of study drug | Censor |
| Baseline tumor assessments only and no evidence of documented PD, treatment discontinuation due to PD or death within no more than one missed visit | Date of 1 <sup>st</sup> dose of study drug | Censor |
| No progression | Date of last visit with adequate assessment | Censor |
| Treatment discontinuation for toxicity or other reason | Date of last visit with adequate assessment | Censor |
| New anticancer treatment started | Date of last visit with adequate assessment | Censor |

Statistical Analysis Plan: Solid Tumor Studies


#### 12.4 Censoring Rules for Overall Survival

| Situation | Date Death or Censoring | Outcome |
|---|---|---|
| Death at any timepoint | Date of death | Death |
| Lost to follow-up immediately after 1 <sup>st</sup><br>dose of study drug | Date of 1 <sup>st</sup> dose study drug | Censored |
| Not known to have died at or after the analysis cutoff date | The date last known alive before data analysis cutoff | Censored |
| Known to have died after the analysis cutoff date | Date of data analysis cutoff | Censored |

Statistical Analysis Plan: Solid Tumor Studies


#### 12.5. Events of Clinical Interest for acalabrutinib

The Events of Clinical Interest (ECIs) have been identified based on preclinical findings, emerging data from clinical studies relating to acalabrutinib, and pharmacological effects of approved BTK inhibitor. The AEs selected for dedicated analysis were evaluated using Standardized MedDRA Queries (SMQs), where available, by SOC, or by Sponsor-defined baskets of MedDRA Adverse Event Grouped Terms.

| Category name | Sub-category name | Definition |
|---|---|---|
| Cardiac events | | SOC Cardiac disorders |
| | Atrial fibrillation | PT Atrial fibrillation PT Atrial flutter |
| Cytopenias –<br>Anemia | | SMQ Haematopoietic erythropenia [narrow + broad] |
| Cytopenias – Leukopenia | | SMQ Haematopoietic leukopenia [narrow + broad] |
| | Neutropenia | <ul> <li>PT Febrile Neutropenia</li> <li>PT Neutropenia</li> <li>PT Neutropenic infection</li> <li>PT Neutropenic sepsis</li> <li>PT Neutrophil count decreased</li> <li>PT Neutrophil percentage decreased</li> </ul> |
| | Other Leukopenia | SMQ Haematopoietic leukopenia [narrow + broad]<br>excluding PTs for neutropenia above |
| Cytopenias -<br>Thrombocytopenia | | SMQ Haematopoietic thrombocytopenia [narrow + broad] |
| Hemorrhage | | SMQ Haemorrhage terms (excl laboratory terms) |
| | Major hemorrhage | As per Acerta definition below |
| Hepatic Events | | <ul> <li>SMQ [narrow] Hepatic failure, fibrosis and cirrhosis and other liver damage-related conditions</li> <li>SMQ [narrow] Liver related investigations signs</li> <li>SMQ [narrow] Hepatitis, non-infectious</li> </ul> |
| Hypertension | | SMQ Hypertension [narrow] |
| Infections | | SOC Infections and infestations |
| Interstitial lung<br>disease/Pneumonitis | | SMQ [narrow] Interstitial lung disease |
| Second primary malignancies | | SMQ Malignant or unspecified tumours and SMQ<br>Myelodysplastic syndrome [narrow] |
| | Second primary malignancies (excluding skin) | SMQ Malignant or unspecified tumours and SMQ<br>Myelodysplastic syndrome [narrow], excluding skin<br>(i.e. exclude SMQ Skin neoplasms, malignant and<br>unspecified) |
| Tumor lysis syndrome | | PT Tumour lysis syndrome |

MedDRA version 20.1

Acerta Pharma 

Statistical Analysis Plan: Solid Tumor Studies


#### **Major Hemorrhage**

Major hemorrhage is defined as any hemorrhagic event that is serious, or Grade ≥ 3 in severity, or that is a central nervous system (CNS) hemorrhage (any severity grade).

#### Search Strategy:

- I. Use standardized MedDRA v19.1 Query:
  - o Haemorrhage terms (excl laboratory terms) (SMQ) [20000039]
- II. Identify Major Events that are a subset of the Haemorrhage SMQ:
  - o Grade > 3 AE
  - o Any SAE
  - o All Grades of CNS hemorrhage

CNS hemorrhage Preferred Terms (MedDRA v19.1):

| CNS hemorrhage Preferred Terms (MedDRA v19.1): | |
|---|---|
| Acute haemorrhagic leukoencephalitis | Haemorrhagic transformation stroke |
| Basal ganglia haematoma | Intracerebral haematoma evacuation |
| Basal ganglia haemorrhage | Intracranial haematoma |
| Basilar artery perforation | Intracranial tumour haemorrhage |
| Brain contusion | Intraventricular haemorrhage |
| Brain stem haematoma | Intraventricular haemorrhage neonatal |
| Brain stem haemorrhage | Meningorrhagia |
| Brain stem microhaemorrhage | Ocular retrobulbar haemorrhage |
| Central nervous system haemorrhage | Optic disc haemorrhage |
| Cerebellar haematoma | Optic nerve sheath haemorrhage |
| Cerebellar haemorrhage | Periventricular haemorrhage neonatal |
| Cerebellar microhaemorrhage | Pituitary haemorrhage |
| Cerebral aneurysm perforation | Putamen haemorrhage |
| Cerebral aneurysm ruptured syphilitic | Ruptured cerebral aneurysm |
| Cerebral arteriovenous malformation haemorrhagic | Spinal cord haematoma |
| Cerebral artery perforation | Spinal cord haemorrhage |
| Cerebral haematoma | Spinal epidural haematoma |
| Cerebral haemorrhage | Spinal epidural haemorrhage |
| Cerebral haemorrhage foetal | Spinal subarachnoid haemorrhage |
| Cerebral haemorrhage neonatal | Spinal subdural haematoma |
| Cerebral microhaemorrhage | Spinal subdural haemorrhage |
| Encephalitis haemorrhagic | Subarachnoid haematoma |
| Epidural haemorrhage | Subarachnoid haemorrhage |
| Extradural haematoma | Subarachnoid haemorrhage neonatal |
| Haemorrhage intracranial | Subdural haematoma |
| Haemorrhagic cerebral infarction | Subdural haematoma evacuation |
| Haemorrhagic stroke | Subdural haemorrhage |
| Subdural haematoma evacuation | Subgaleal haematoma |
| Subdural haemorrhage | Thalamus haemorrhage |
| Subdural haemorrhage neonatal | Traumatic intracranial haemorrhage |

Acerta Pharma 

Statistical Analysis Plan: Solid Tumor Studies


### 12.6. Events of Clinical Interest for a combination of acalabrutinib and pembrolizumab

The Events of Clinical Interest (ECIs) for a combination treatment have been identified based on preclinical findings, emerging data from clinical studies, and finding from post marketing (for pembrolizumab).

The AEs selected for dedicated analysis were evaluated using Standardized MedDRA Queries (SMQs), where available, by SOC, by PT or by Sponsor-defined baskets of MedDRA Adverse Event Grouped Terms.

| Category name | Sub-category name | Definition |
|---|---|---|
| Cytopenias – | | SMQ Haematopoietic erythropenia [narrow + |
| Anemia | | broad] |
| Cytopenias – Leukopenia | | SMQ Haematopoietic leukopenia [narrow + broad] |
| | Neutropenia | <ul> <li>PT Febrile Neutropenia</li> <li>PT Neutropenia</li> <li>PT Neutropenic infection</li> <li>PT Neutropenic sepsis</li> <li>PT Neutrophil count decreased</li> <li>PT Neutrophil percentage decreased</li> </ul> |
| | Other Leukopenia | SMQ Haematopoietic leukopenia [narrow + broad]<br>excluding PTs for neutropenia above |
| Infections | | SOC Infections and infestations |
| Transaminases elevation | | <ul> <li>PT Alanine aminotransferase increased</li> <li>PT Aspartate aminotransferase increased</li> <li>PT Transaminases increased</li> </ul> |
| Immune-mediated pneumonitis | | PT Pneumonitis |
| Immune-mediated colitis | | PT Colitis |
| Immune-mediated hepatitis | | <ul><li>PT Hepatitis</li><li>PT Autoimmune hepatitis</li></ul> |
| Immune-mediated<br>endocrinopathies -<br>Hypophysitis | | <ul><li>PT Hypophysitis</li><li>PT Hypopituitarism</li><li>PT Adrenal insufficiency</li></ul> |
| Immune-mediated endocrinopathies - Thyroid disorders | | <ul><li>PT Hyperthyroidism</li><li>PT Hypothyroidism</li><li>PT Thyroiditis</li></ul> |
| Immune-mediated endocrinopathies - Type 1 diabetes | | <ul><li>PT Type 1 diabetes mellitus</li><li>PT Diabetic ketoacidosis</li></ul> |
| Immune-mediated nephritis | | PT Nephritis |
| Immune-mediated skin adverse reactions | | <ul><li>PT Stevens-Johnson syndrome</li><li>PT Toxic epidermal necrolysis</li></ul> |

MedDRA version 20.1

Acerta Pharma 